CLINICAL TRIAL: NCT05782205
Title: Surgeons' Mental Distress and Risks After Severe Complications Following Radical Gastrectomy in China: a Nationwide Cross-Sectional Questionnaire
Brief Title: Surgeons' Mental Distress and Risks After Severe Complications Following Radical Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, hongyong he, Clinical Professor, Shanghai Zhongshan Hospital
Other Study IDs: Zhongshan-HHY-01
Record Dates: First submitted 2023-03-09; First posted 2023-03-23 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Severe complications following radical gastrectomy — The respondents are limited to surgeons who had previously experienced severe complications following radical gastrectomy as chief surgeons.

SUMMARY:
Surgeons experience higher levels of work stress, even under normal circumstances. Many can suffer from substantial levels of mental health issues, especially when faced with severe complications. However, due to a variety of reasons, many surgeons are reluctant to disclose mental health issues or seek psychological help.

Gastric cancer is the fifth most common malignancy globally and accounts for the fourth leading cause of death from cancer. In China specifically, gastric cancer is a major public health issue, with some 400,000 new cases diagnosed every year. Of those cases, more than 80% patients are at advanced stages when diagnosed. At present, radical gastrectomy is considered the standard approach for patients with resectable advanced gastric cancer. Severe complications following radical gastrectomy ranged from 2.7% to 9.4% worldwide. In addition to delaying patients' recovery courses, severe complications also place enormous pressure on chief surgeons who performed the operations. Such pressures may bring great risks of psychological distress.

Surgeons are also the victims when they encounter severe complications following radical gastrectomy. Their mental distress should not be minimized. Until now, little has been known about the effects of surgical complications on surgeons. In the current study, based on a large-scale questionnaire survey in China, the investigators aimed to investigate incidences of surgeons' mental distress following severe complications after radical gastrectomy. The investigators also aimed to identify independent risk factors which could help develop strategies to improve the mental well-being of these surgeons after such incidences.

ELIGIBILITY:
Inclusion Criteria:

* General and/or gastrointestinal surgeons who experienced severe complications after radical gastrectomy.

Exclusion Criteria:

* Other conditions that do not meet the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Enrolled as many surgeons as possible within the research time
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Surgeons' mental health | June 01, 2023 to August 31, 2024.
  The clinical features collected in the questionnaire relating to the surgeons' mental distress included: i) feeling burnout, anxiety, or depression; ii) avoiding radical gastrectomy or feeling stress, slowing down the process during radical gastrectomy operations; iii) having physical reactions, including heart pounding, trouble breathing, or sweating while recalling; iv) having urges to quit being a surgeon; v) taking psychiatric medications; and vi) seeking psychological counseling. Meeting any one of the above six clinical features was regarded as having mental distress; Meeting ore or two was defined as mild mental distress, and meeting three or more was defined as severe mental distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He H, Lin C, Li R, Zang L, Huang X, Liu F. Surgeons' mental distress and risks after severe complications following radical gastrectomy in China: a nationwide cross-sectional questionnaire. Int J Surg. 2023 Aug 1;109(8):2179-2184. doi: 10.1097/JS9.0000000000000463. PMID 37158145